CLINICAL TRIAL: NCT05273567
Title: A Randomized Controlled Trial of Guanfacine-er for Cannabis Use Disorder
Brief Title: A Trial of Guanfacine-er for Cannabis Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christina Ann Brezing, Assistant Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8103; 1K23DA045080-01A1 (NIH)
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Cannabis Use
Keywords: cannabis; guanfacine; treatment
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Guanfacine-ER (Experimental): Participants will start on guanfacine-ER 1mg nightly for 1-week (week 1) and slowly increase by 1mg/per week to a max dose of 4mg per day or maximum dose as tolerated. Medication taper to discontinuation will begin in week 11 and continue into week 12 until complete by end of study, decreasing the dose by 1mg every 4 days until stopped.
  Interventions: Drug: guanfacine-ER
- Placebo (Placebo Comparator): Placebo will be taken nightly and titrated and tapered similar to the active arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: guanfacine-ER — guanfacine-er dispensed daily, starting at 1mg and increasing to 4mg/day or the maximum tolerated dose.
  Other Names: Intuniv-er
  Arms: Guanfacine-ER
Other: Placebo — placebo will be dispensed similar to the active arm.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to investigate the effect of guanfacine-ER on reductions in cannabis use and explore its effects on impulsivity and withdrawal through a hybrid in-person and virtual trial of treatment-seeking individuals with Cannabis Use Disorder (CUD), and assessing the feasibility of the virtual components of the study.

DETAILED DESCRIPTION:
This will be a 12-week randomized, double-blind, placebo-controlled trial, of guanfacine-ER compared to placebo for CUD. Participants will start on guanfacine-ER 1mg nightly for 1-week (week 1) and slowly increase by 1mg/per week to a max dose of 4mg or maximum dose as tolerated through week 4. Patients will be maintained on the medication through week 11. During week 11, they will begin a taper to discontinuation, decreasing the dose of guanfacine by 1mg every 4 days until stopped during the last week of the study (week 12). The primary purpose of this study is therefore to investigate the effect of guanfacine-ER on reductions in cannabis use and explore its effects on impulsivity and withdrawal through a hybrid in person and virtual trial of treatment-seeking individuals with CUD. In light of COVID-19 viral transmission mitigation policies, we will make use of the technological applications of virtual visits, remote administration of urine drug testing and medication, and ecological momentary assessments (EMA) in conjunction with once monthly in person visits to the clinic during weeks 1, 4, 8, 12.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-V criteria for a current cannabis use disorder
* Seeking treatment for cannabis use disorder with goal to reduce or stop use
* THC-positive drug screen
* Capable of giving informed consent and complying with study procedures
* Access to internet and devices capable of completing study procedures
* capability of receiving mailed packages for study supplies

Exclusion Criteria:

* Lifetime history of DSM-V diagnosis of schizophrenia or schizoaffective disorder
* Current DSM-V criteria for a psychiatric disorder supported by the MINI that in the investigator's judgment is unstable, would be disrupted by the study medication, or is likely to require new pharmacotherapy or psychotherapy during the study period. Individuals who are currently stable on psychotropic medication for at least 2 months may be included if in the investigator's opinion the psychotropic medication is compatible with the study medication (guanfacine-ER). Any medical or psychiatric conditions that in the investigator's judgment would interfere with safe participation in the study will be exclusionary.
* Individuals who meet DSM-V criteria for any moderate to severe substance use disorder other cannabis, caffeine or nicotine use disorders
* Pregnancy, lactation, or failure to use adequate contraceptive method in female patients who are currently engaging in sexual activity that can result in pregnancy
* Legally mandated to participate in a substance use disorder treatment program
* Current or recent history of significant violent or suicidal behavior, risk for suicide or homicide
* Known history of allergy, intolerance, or hypersensitivity to guanfacine
* Bradycardia (< 50 beats/minute), hypotension (sitting or standing BP < 90/50), or symptoms attributable to hypotension (i.e. lightheadedness or dizziness on standing)
* Individuals currently being treated with the antihypertensive medications, including the class of alpha 2 agonists that have a potential drug-interaction with guanfacine based on adrenergic modulation
* Individuals currently taking medications that may interact adversely with guanfacine and deemed not clinically safe by study physician at consent, such as rifampicin, ketoconazole, St. John's Wort, and amitriptyline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change in daily cannabis use as measured by ecological momentary assessments (EMA). | 12 weeks of study
  Change in number of days of use per week as compared to baseline. Participants will complete ecological momentary assessments (EMA) daily on any internet-accessible device (smart phone, computer, tablet). The daily EMA will assess cannabis use during quartiles of the day. Participants will mark "Yes" if they used cannabis from 12AM-6AM, 6AM-12PM, 12PM-6PM, or 6PM-12AM for each 24 hour period of the study. Primary Outcome will dichotomize each day as a use day (1) or a non using day (0).

CONTACTS AND LOCATIONS:
Overall Officials: Christina Brezing, MD, Principal Investigator — NYSPI
Locations (1):
- STARS Clinic at Columbia and NYSPI Department of Psychiatry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results published in this report (after de-identification) (text, tables, figures)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: beginning twelve months and ending 5 years after article publication
Access Criteria: to researcher who provides a methodologically sound proposal to achieve aims in approved proposal